CLINICAL TRIAL: NCT04925089
Title: Pilot Study of ctDNA and Imaging Characteristics as Biomarkers of Disease-related Outcomes in Patients With Localized Leiomyosarcoma Receiving Chemotherapy
Brief Title: Localized Leiomyosarcoma Biomarker Protocol
Status: Recruiting | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HUM00219057; HUM00213723 (Other: University of Michigan); 1P50CA272170-01 (NIH)
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Leiomyosarcoma
Keywords: ctDNA; radiomics; biomarker
MeSH Terms: conditions — Leiomyosarcoma | interventions — Blood Specimen Collection; Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be obtained after enrollment for analysis of germ-line DNA and for ctDNA. Archival tissue will be collected and analyzed for gene mutations in leiomyosarcoma. Tumor tissue from sarcoma resection will be collected and analyzed for genetic changes in leiomyosarcoma after treatment. Digital Images will be collected and analyzed for change in imaging characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and Tissue collection — Blood and tissue will be collected and analyzed for detection of ctDNA and genetic change

SUMMARY:
* Leiomyosarcoma (LMS) is one of the more common soft tissue sarcomas (STS).
* Patients presenting with large, high-grade, localized LMS are at significant risk of developing metastasis following curative surgery.
* Clinical trials of neoadjuvant or adjuvant anthracycline and ifosfamide have suggested that patients with localized STS who are at high-risk of metastasis may benefit from chemotherapy, but the magnitude of benefit in unselected patient population is relatively small.
* Currently, patient age, and tumor size and grade are used to assess risk of metastases and survival
* Studies evaluating tumor response by imaging and histopathology have not established correlation between tumor characteristics as biomarkers for risk of metastasis or sarcoma recurrence.
* Circulating tumor DNA (ctDNA) is present in blood of patients with advanced/metastatic LMS and may serve as biomarker of tumor response to chemotherapy. Blood samples will be collected prior to, during and after chemotherapy and analyzed for ctDNA and for mutations in genes that are associated with increased risk of developing sarcoma. Tumor tissue will be collected and analyzed for changes in genes. Digital images of the sarcoma from CT or MRI scans obtained during treatment will be obtained for advanced radiomic analysis. Patients will be followed for 2 years after study entry for signs of sarcoma recurrence.
* A biomarker of tumor response and patient survival benefit from chemotherapy early in the course of chemotherapy would be of significant impact in treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized leiomyosarcoma (LMS) of extremity, body wall or retroperitoneum
* Grade 2 or 3, or high-grade LMS
* Tumor size >5 cm in greatest dimension
* Primary tumor amenable to complete resection
* There is no age requirement
* Participant agrees to receive neoadjuvant doxorubicin and ifosfamide combination chemotherapy
* If pre-operative radiation is administered, it must be administered after chemotherapy. Post-operative radiation may be administered
* Archival tumor tissue (either frozen sample, tissue block containing tumor, or minimum of 4 unstained slides and 1 H&E stained slide) from diagnostic or pre-treatment biopsy available for study research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been diagnosed with grade 2 or 3, high-grade leiomyosarcoma who have agreed to receive neoadjuvant doxorubicin and ifosfamide combination chemotherapy where the primary tumor is amenable to complete resection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the association between tumor characteristics assessed by contrast-enhanced MRI and location with presence of circulating tumor DNA (ctDNA) in patients with localized, high-grade leiomyosarcoma | 2 years
  Tumor characteristics from imaging will be compared to the presence of circulating tumor DNA , obtained from blood samples over multiple time points
To evaluate change in ctDNA in patients with localized, high-grade leiomyosarcoma undergoing preoperative doxorubicin/ifosfamide chemotherapy with or without pre-operative radiation | 2 years
  Blood will be collected at multiple timepoints. The presence of ctDNA will be assessed prior to, during, and after treatment with chemotherapy and / or radiation

SECONDARY OUTCOMES:
To examine the association of change in ctDNA and imaging characteristics with 2-year relapse-free survival | 2 years
  The change in the presence of ctDNA from serial blood collection will be compared to the absence of sarcoma recurrence or after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, Principal Investigator — University of Michigan Rogal Cancer Center
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
We will share deidentified genetic data on the NIH site, and deidentified imaging data will be shared with the lab at Columbia University. We are not sharing patient identities.

REFERENCES:
- [Derived] Kasper B, Wilky BA. Sounding the Alarm on Leiomyosarcoma Recurrence: Role of Circulating Tumor DNA. Clin Cancer Res. 2022 Jun 13;28(12):2480-2481. doi: 10.1158/1078-0432.CCR-22-0738. PMID 35412607